CLINICAL TRIAL: NCT00091468
Title: Double-Blind Treatment of Mild Cognitive Impairment (MCI) With Transdermal Nicotine or Transdermal Placebo
Brief Title: Nicotine Treatment of Mild Cognitive Impairment (MCI)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Paul Newhouse, M.D., University of Vermont
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IA0060; R01AG022462-02 (NIH)
Record Dates: First submitted 2004-09-09; First posted 2004-10-14 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Age-Related Memory Disorders
Keywords: Age-Related Memory Loss; Nicotine; Mild Cognitive Impairment (MCI)
MeSH Terms: conditions — Memory Disorders; Cognitive Dysfunction | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Group (Placebo Comparator): Placebo for first six months of study; moved to open-label active nicotine for second six months
  Interventions: Drug: Placebo transdermal patch
- Active Nicotine Group (Experimental): Blinded active nicotine for first six months of study; open-label active nicotine for second six months
  Interventions: Drug: Transdermal nicotine patch

INTERVENTIONS:
Drug: Transdermal nicotine patch — double-blind phase: 5mg for 1 week, 10mg for 2 weeks, 15mg for 23 weeks open label phase: 5mg for 1 week, 10mg. for 2 weeks, 15mg. for 23 weeks taper down: 10mg. for 2 weeks, 5mg. for 1 week
  Other Names: Nicotrol
  Arms: Active Nicotine Group
Drug: Placebo transdermal patch — placebo patch, 5mg for 1 week, 10mg for 2 weeks, 15mg for 23 weeks
  Arms: Placebo Group

SUMMARY:
The purpose of this 12-month study is to determine whether nicotine, administered in the form of nicotine patches, can improve symptoms of memory loss in some people experiencing mild memory problems (referred to in this study as "mild cognitive impairment" or MCI).

DETAILED DESCRIPTION:
The purpose of this study is to determine whether nicotine can improve symptoms of memory loss in some people experiencing mild memory problems (referred to in this study as "mild cognitive impairment" or MCI). The study will last approximately 12 months and will be conducted at 3 clinical sites in the United States.

Recent studies have suggested that one of the causes of memory disorders may be a reduction in a particular chemical substance in the brain. This chemical substance, acetylcholine, is thought to act on certain brain cells in a specific way that helps us to remember and use memories as well as affect our mood. In MCI (and Alzheimer's disease), the level of acetylcholine may be changed, and this may impair brain functioning. Preliminary studies have suggested that short-term administration of nicotine appears to improve memory in patients with mild memory loss and early Alzheimer's disease. Nicotine imitates many of the actions of acetylcholine. By administering nicotine over a longer period of time to patients with MCI, this study could lead to a better understanding of whether nicotine can act to improve memory loss symptoms over the longer term and whether it can help delay the progression of memory loss symptoms. The amount of nicotine in each patch used in this study is the same level found in patches that are used in people who are trying to quit smoking.

This study will include up to twelve visits.

ELIGIBILITY:
Specific Inclusion Criteria:

* Age 55+.
* Memory complaints and memory difficulties which are verified by an informant.
* Abnormal memory function documented by scoring below the education adjusted cutoff on the Logical Memory II subscale (Delayed Paragraph Recall) from the Wechsler Memory Scale - Revised (the maximum score is 25):

  1. less than or equal to 8 for 16 or more years of education,
  2. less than or equal to 4 for 8 - 15 years of education,
  3. less than or equal to 2 for 0 - 7 years of education.
* Mini-Mental Status Exam score between 24 and 30 (inclusive).
* Clinical Dementia Rating of 0.5 with a memory box score of 0.5 or 1.0.
* General cognition and functional performance sufficiently preserved such that a diagnosis of Alzheimer's disease cannot be made by the site physician at the time of the screening visit.
* No significant cerebrovascular disease: Modified Hachinski score of less than or equal to 4.
* Stable medications for at least 1 month prior to screening.
* Hamilton Depression rating scale score of less than or equal to 12 on the 17-item scale.
* Informant is available who has frequent contact with the participant (e.g. an average of 10 hours per week or more).
* Adequate visual and auditory acuity to allow neuropsychological testing.
* Good general health with no additional diseases expected to interfere with the study.
* Any conditions that subject may have must be stable for 3 months prior to screening.
* Participant is not pregnant, lactating, or of childbearing potential (i.e. women must be two years post-menopausal or surgically sterile).
* Participants will be taking no drugs with pro- or anti-cholinergic properties.

Exclusion Criteria:

* Any significant neurologic disease such as Alzheimer's disease, Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic deficits or known structural brain abnormalities.
* Major depression or another major psychiatric disorder as described in DSM-IV within the past 2 years.
* History of alcohol or substance abuse or dependence within the past 2 years (DSM IV criteria).
* Any significant, unstable medical condition.
* Use of any investigational drugs within 30 days or 5 half-lives, whichever is longer, prior to screening.
* Any tobacco use within the past year.

Exceptions to these specific Inclusion and Exclusion Criteria (e.g., WMS-R cutoffs) may be made on a case by case basis by the Principal Investigator.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2003-09; Primary Completion 2008-07 (Estimated); Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
Safety of transdermal nicotine patch | 13 months

SECONDARY OUTCOMES:
Change in cognitive performance | 13 months
Change in global functioning | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Newhouse, MD, Principal Investigator — University of Vermont
Locations (3):
- United States (3):
  - Georgetown University Medical Center, Department of Neurology, Washington D.C., District of Columbia
  - Duke University, Duke Health Center at Morreene Road, Durham, North Carolina
  - University of Vermont College of Medicine, Burlington, Vermont

REFERENCES:
- [Background] Newhouse PA, Potter A, Singh A. Effects of nicotinic stimulation on cognitive performance. Curr Opin Pharmacol. 2004 Feb;4(1):36-46. doi: 10.1016/j.coph.2003.11.001. PMID 15018837
- [Background] Newhouse P, Singh A, Potter A. Nicotine and nicotinic receptor involvement in neuropsychiatric disorders. Curr Top Med Chem. 2004;4(3):267-82. doi: 10.2174/1568026043451401. PMID 14754447
- [Background] Newhouse PA, Potter A, Kelton M, Corwin J. Nicotinic treatment of Alzheimer's disease. Biol Psychiatry. 2001 Feb 1;49(3):268-78. doi: 10.1016/s0006-3223(00)01069-6. No abstract available. PMID 11230878
- See also: Nicotine Treatment of Mild Cognitive Impairment (MCI) study at University of Vermont — http://www.uvm.edu/~cnru/